CLINICAL TRIAL: NCT03415334
Title: Use of Public Health Approaches for HCV Elimination in an Egyptian Model Village
Brief Title: Effect of Implementation Of Outreach Behavioral Change Program for HCV Elimination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre, Egypt (Other)
Collaborators: Egyptian Liver Hospital (Other)
Responsible Party: Principal Investigator, Prof.Dr. Ammal Mokhtar Metwally, Head of community medicine research department, National Research Centre, Egypt
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 66187
Record Dates: First submitted 2018-01-13; First posted 2018-01-30 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Hepatitis C and B VIRUS Screening, Awareness and Behavior Assessment and Evaluation for All Inhabitants Above Twelve Years of Al Othmaneya Village
Keywords: Hepatitis C; social marketing; Communication for behavior development
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Intervention Model Description: The study passed through three phases; first phase pre-interventional assessment of level of the recommended behavior development towards eradication of HCV, dominance of current risky behaviors and the wrong believes regarding HCV . The second phase included: community based interventions and the setting of the educational activation plan for HCV elimination in the village and the third was post-intervention evaluation of the change of level of community behaviors adoption according to a preset indicators.
Masking Description: care providers were not the same persons who did the assessment and the evaluation .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- behavioral change (Other): two approaches for behavior changes : social marketing and behavioral development
  Interventions: Behavioral: behavioral development for change

INTERVENTIONS:
Behavioral: behavioral development for change — 1. Social Marketing Principles (4 Ps) Product, price, place and promotion
  2. Communication for Behavior Development Approach 1. Interpersonal communication campaigns (IPC) 2. Mass media and public gathering awareness campaigns 3. Public health awareness campaigns 4. A village hotline and local satellite channel 5. School awareness raising events
  Other Names: 2 approaches were used : 1) Social Marketing Principles (4Ps) 2) Communication for Behavior Development Approach

SUMMARY:
Elimination of hepatitis C virus (HCV) is the process of stopping sustained transmission of viral hepatitis, reducing its incidence to zero and providing access to safe, affordable and effective treatment and care for everyone. Consequently, HCV will not be a leading cause of mortality (1). The World Health Organization (WHO) called for comprehensive programs that enhance access to affordable treatment in developing countries as HCV was considered a global public health priority since 2010 and set criteria of elimination(2). A disease is eliminated if its controlling efforts are sufficient to prevent an epidemic from occurring in a given geographical area and measures must be continued to prevent re-establishment of transmission (3) According to the Centers for Disease Control and Prevention (CDC), HCV now surpasses HIV as the nation's deadliest blood-borne disease. In addition, the majority of infected persons are not aware of their infection as they are not clinically ill and there is no vaccine for Hepatitis C. It is well known that the best way to prevent Hepatitis C is by avoiding behaviors that can spread the disease. (4) This study is a way forward for the elimination of hepatitis C from Egypt through applying different public health approaches for motivating people and changing villagers' risky behaviors aiming at increasing the number of people adopting healthy practices for decreasing the incidence rate of hepatitis in El Othmaneya village. The proposed activities along one year were applied for 3575 inhabitants aged more than 12 years who were get tested for Hepatitis C Virus (HCV) antibodies. The initiative activities were provided by community-led coalition and supported technically by the Egyptian Liver Research Institute and Hospital (ELRIAH).

DETAILED DESCRIPTION:
The objective of the outreach village initiative is to capture in more detail the dominance of the risky behaviors as well as the level of behavior development and putting adaptive motivational strategies aiming at behavior change. In addition, the initiative set public health approaches for HCV elimination and evaluate its efficacy in changing behaviors.

Methodology The initiative was interventional evaluation study which was conducted along 24 months starting from May 2015 to October 2017.

Phases of the study:

The study passed through three phases; first phase pre-interventional assessment of level of the recommended behavior development towards eradication of HCV, dominance of current risky behaviors and the wrong believes regarding HCV . The second phase included: community based interventions and the setting of the educational activation plan for HCV elimination in the village and the third was post-intervention evaluation of the change of level of community behaviors adoption according to a preset indicators.

Indicators are the following:

Awareness:

1. Using previously used syringes
2. Sharing shaving equipment, nail cutters or through needle stick injury
3. Defect in infection control process during sessions for teeth treatment
4. sharing tooth brush with other family members
5. It is better for HCV patients to get vaccinated with Hepatitis B vaccines
6. Using new syringes/sharp instruments which are not used before could reduce the risk of becoming infected with HCV
7. Awareness by the recommended behaviors can limit the complication and propagation of HCV infection

Perception:

1. HCV is a serious disease
2. Hepatocellular carcinoma (HCC) is a complication of HCV
3. Cirrhosis is a complication of HCV
4. Early diagnosis could make a change in patients' health
5. Fatigue from least effort is symptom of HCV

The Attitude:

1. Asking the barber: to change the shaving tools in front of them
2. to use their own shaving machine
3. Checking for sterilized tools at dentist clinic
4. Telling the dentist if they have/ had HCV

The tried out / rejected or adopted : Not sharing:

1. nail cutters and scissors between family members
2. loofah and sponge for personal cleaning
3. the use of scarves' pins by the veiled females in the same family
4. other's shaving tools
5. others tooth brushes

ELIGIBILITY:
Inclusion Criteria:

All village inhabitants starting from 12 years old

Exclusion Criteria:

inhabitants less than 12 years old

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3575 (Actual)
Dates: Start 2015-05-21 (Actual); Primary Completion 2017-05-13 (Actual); Study Completion 2017-10-21 (Actual)

PRIMARY OUTCOMES:
percent change of awareness using pre and post intervention questionnaire for participants who became aware of the problem | two years
  1. Using previously used syringes
  2. Sharing shaving equipment, nail cutters or through needle stick injury
  3. Defect in infection control process during sessions for teeth treatment
  4. sharing tooth brush with other family members
  5. It is better for HCV patients to get vaccinated with Hepatitis B vaccines
  6. Using new syringes/sharp instruments which are not used before could reduce the risk of becoming infected with HCV
  7. Awareness by the recommended behaviors can limit the complication and propagation of HCV infection
Percent change using pre and post intervention questionnaire for participants who became concerned about the problem,acquired knowledge and internalized the knowledge | two years
  Perception:
  1. HCV is a serious disease
  2. HCC is a complication of HCV
  3. Cirrhosis is a complication of HCV
  4. Early diagnosis could make a change in patients' health
  5. Fatigue from least effort is symptom of HCV
Percent change using pre and post intervention questionnaire for participants who became motivated and had positive attitude to do something about the problem | two years
  The Attitude:
  1. Asking the barber: to change the shaving tools in front of them
  2. to use their own shaving machine
  3. Checking for sterilized tools at dentist clinic
  4. Telling the dentist if they have/ had HCV
Percent change of behavior using pre and post intervention questionnaire for participants who tried out /rejected or adopted the recommended behavior | two tears
  The tried out / rejected or adopted : Not sharing:
  1. nail cutters and scissors between family members
  2. loofah and sponge for personal cleaning
  3. the use of scarves' pins by the veiled females in the same family
  4. other's shaving tools
  5. others tooth brushes

IPD SHARING:
Plan to Share IPD: Undecided
After Approval of clinical Trial.gov and having ID

REFERENCES:
- [Background] Barrett S. Eradication versus control: the economics of global infectious disease policies. Bull World Health Organ. 2004 Sep;82(9):683-8. PMID 15628206
- [Background] 4) Center for Disease Control (CDC). Division of Viral Hepatitis (DVH) Strategic Plan, 2016-2020: Bringing Together Science and Public-Health Practices for the Elimination of Viral Hepatitis. (2016). http://www.cdc.gov/hepatitis/pdfs/dvh-strategicplan2016-2020-draft.
- [Background] WORLD HEPATITIS SUMMIT HARNESSES GLOBAL MOMENTUM TO ELIMINATE VIRAL HEPATITIS. Cent Eur J Public Health. 2015 Sep;23(3):272. No abstract available. PMID 26618210
- [Background] Heymann DL. Control, elimination, eradication and re-emergence of infectious diseases: getting the message right. Bull World Health Organ. 2006 Feb;84(2):82. doi: 10.2471/blt.05.029512. Epub 2006 Feb 23. No abstract available. PMID 16501719
- See also: Related Info — https://l.facebook.com/l.php?u=https%3A%2F%2Fwww.surveymonkey.com%2Fr%2Fbe3ha6vio8r&h=ATN51FLS53cw_g64r8dtnrqdze4aVvqchGW--CsmYwVFbCA3OZCUL34Ke2HqSSCCvzEjD7V0zEd2YRogu0dYlMKvWqJFRO_dfovM35_zMNACDYbuovdU6kBHdypVWRzM7B4tsDl3nA&s=1&enc=AZOZGroIjCOtl-PbtUSzPfc_zbXXrXIl4aXi4MU1mRHtUAJEhnvdVxHCQ2OlfPy8UA9nmlb0FPGnP8fIi4ATLYQO
- See also: Related Info — http://www.liver-ri.org.eg/en/towards-a-village-free-from-hepatitis/about-towards-a-village-free-from-hepatitis-project